CLINICAL TRIAL: NCT01535495
Title: Propranolol for Diabetic Retinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 2011-0475
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: beta-antagonist; propranolol; diabetic retinopathy; diabetes; angiogenesis; neovascularization
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Neovascularization, Pathologic | interventions — Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Complete laser (Experimental): Patients who have had complete panretinal photocoagulation laser treatment and active retinal neovascularization
  Interventions: Drug: Propranolol
- Laser naive (Experimental): Patients who have not had panretinal photocoagulation laser treatment and active retinal neovascularization without so called "high-risk" characteristics
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — Propranolol XL 120mg by mouth once daily
  Other Names: Both groups receive the same intervention

SUMMARY:
This study is investigating if the oral beta antagonist propranolol can induce regression of retinal neovascularization associated with proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
Oral propranolol 120mg daily will be given to 10 patients with proliferative diabetic retinopathy over a 12 week period to evaluate the effect on retinal neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years
* Eyes with proliferative diabetic retinopathy and neovascularization
* Eyes with a history of panretinal photocoagulation treatment and persistent neovascularization deemed by the investigator to be a potential threat to visual acuity either by causing a vitreous hemorrhage or tractional retinal detachment. (Group 1 - maximum 5 eyes enrolled with these characteristics)
* Eyes without a history of panretinal photocoagulation treatment, but that do not have high-risk proliferative diabetic retinopathy characteristics (i.e. these are eyes that have early proliferative diabetic retinopathy that are not yet at a high-risk for vitreous hemorrhage and tractional retinal detachment such that panretinal photocoagulation laser may be deferred). (Group 2 - maximum 5 eyes enrolled with these characteristics)

Exclusion Criteria:

* Either panretinal photocoagulation laser or focal/grid laser into study eye within 3 months of study enrollment
* Anti-Vascular endothelial growth factor injection into study eye within 3 months of study enrollment
* Contraindications to beta-blockers such as: allergy, previous intolerance, abnormally slow heart rates, asthma or chronic obstructive pulmonary disease, use of medications that have an effect on certain drug metabolic pathways that may cause interactions.
* Known coronary arterial disease or left ventricular dysfunction, or known peripheral vascular disease
* Resting heart rate <60 or systolic blood pressure <90 and/or diastolic blood pressure <50
* Pregnancy
* All patients will either be post-menopausal, have adequate birth control and, if of childbearing age, will have a urinary pregnancy test performed
* Allergy to fluorescein dye
* Media opacity obscuring adequate determination of neovascularization including dense cataract or dense vitreous hemorrhage
* Patient is already taking an oral beta-blocker
* Vulnerable populations such as prisoners and minors will also be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Area of retinal neovascularization on fundus photography | 12 weeks

SECONDARY OUTCOMES:
Retinopathy level in contralateral eye | 12 weeks
Optical coherence tomography macular thickness of treated and fellow eye | 12 weeks
Amount of fluorescein leakage on angiography | 12 weeks
Early Treatment Diabetic Retinopathy Study visual acuity in study and fellow eye | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Ip, MD, Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States